CLINICAL TRIAL: NCT07034053
Title: Clofarabine Therapy in Patients With Locally Advanced or Metastatic Urothelial Carcinoma: a Phase 1/2 Dose-Escalation Study
Brief Title: Clofarabine Therapy in Locally Advanced or Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ekaterina Laukhtina (Other)
Responsible Party: Sponsor-Investigator, Ekaterina Laukhtina, Dr. Sponsor-Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOFARABINE_UC
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Advanced Urothelial Carcinoma; Metastatic Urothelial Cancer
MeSH Terms: interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with urothelial carcinoma treated with clofarabine (Experimental)
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Patients receive i.v. clofarabine in a dose-escalation regimen

SUMMARY:
This phase 1/2 study will evaluate the maximum tolerated dose, efficacy, and safety of clofarabine in patients with advanced or metastatic urothelial cancer.

DETAILED DESCRIPTION:
Clofarabine is an antimetabolite chemotherapeutic agent used as a subsequent line of treatment in pediatric patients with leukemia. In preclinical studies, it showed promising results, surpassing the effectiveness of the current standard of care. The study aims to define the maximum tolerated dose of clofarabine in patients with metastatic or locally advanced urothelial carcinoma. It also seeks to characterize the pharmacokinetics of clofarabine and assess the efficacy, safety, and tolerability of the treatment. The study population consists of patients with histologically confirmed urothelial carcinoma and radiologically documented metastatic or unresectable locally advanced disease, who have already received standard-of-care treatment. The study will be performed using a dose-escalation regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed urothelial carcinoma, radiologically documented metastatic or unresectable locally advanced disease
* Patients who have already received standard treatment and did not benefit from it, or patients who have refused standard therapy
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) greater than or equal to 1500.
* White blood cell (WBC) count greater than 3.0.
* Platelets greater than or equal to 100.
* Hemoglobin greater than 9.0 g/dL.
* Adequate hepatobiliary function as indicated by the following laboratory values: Total bilirubin ≤ 1.5 x upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Adequate renal function as indicated by the following laboratory values: Serum creatinine ≤ 1.0 mg/dL; if serum creatinine > 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease (MDRD) equation
* Adequate cardiac function (NYHA cardiac III-IV excluded)
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Willing and able to provide informed consent

Exclusion Criteria:

* Received previous treatment with clofarabine
* Current concomitant chemotherapy, radiation therapy, or immunotherapy
* Prior radiation therapy to the pelvis
* Currently participation in other investigational drug studies or having received other investigational drugs within the previous 30 days
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment. In particular: a) New York Heart Association classification stage II, III, or IV congestive heart failure; b) Coronary artery disease or arteriosclerotic cardiovascular disease (angina, myocardial infraction) within 3 months of first dose of study drug; c) Any other primary cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Any medical condition that requires chronic use of oral high-dose corticosteroids (in excess of 1 mg/kg/day) (low-dose corticosteroid for pre-medication purposes are allowed).
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Diagnosis of another malignancy, unless the patient has been disease-free for at least 5 years following the completion of curative intent therapy with the following exceptions: Patients with treated non-melanoma skin cancer, in-situ carcinoma or cervical intraepithelial neoplasia regardless of disease-free duration are eligible for this study if definitive treatment for the condition has been completed; Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on PSA value are eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed
* Had currently active gastrointestinal disease, or prior surgery that might affect the ability of the participants to absorb oral Clofarabine.
* Had prior treatment with a known nephrotoxic drug within 2 weeks of the first dose of study drug, unless the participants had a calculated GFR >30 at 2 time points no <7 days apart during the 2- week period prior to the first dose of study drug.
* Positive human immunodeficiency virus (HIV) test.
* Female patients who are pregnant/breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Determining the maximum tolerated dose (MTD) | From the start of study drug administration through the first 28 days of dosing (Cycle 1), based on the observed incidence of dose-limiting toxicity (DLT) and evaluation of maximum tolerated dose (MTD)
  The objective of the dose selection phase is to determine the maximum tolerated dose (MTD) or confirm that the start dose level of clofarabine is safe. The MTD is defined as the highest dose at which the probability of toxicity remains below the target toxicity threshold. MTD estimation will be based on the observed dose-dependent incidence rate of dose-limiting toxicity (DLT) within the first 28 days of dosing (Cycle 1).
  Patients eligible for MTD evaluation include:
  * Those who completed Cycle 1 and took at least 80% of the required total dose of the study drug (protocol-defined dose reductions will not be considered noncompliance).
  * Those who discontinued during Cycle 1 due to a DLT.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From the date of study treatment start until the date of the best documented objective response (for a maximum duration of 36 months).
  Objective response rate (ORR) is defined as the percentage of patients whose best response is either a complete response (CR) or partial response (PR). Patients for whom best tumor response is not CR or PR, as well as patients without any efficacy assessment will be considered non-responders. According to RECIST v1.1, confirmation of PR and CR is not required considering the nature of the study and the protocol requirements.
Duration of response (DOR) | From the date of the first documented objective response of PR or CR, whichever is noted earlier, to disease progression or death (for a maximum duration of 36 months).
  Duration of response (DOR) (for PR and CR) is defined as the time from the first documented objective response of PR or CR, whichever is noted earlier, to disease progression or death (if death occurs before progression is documented). DOR will be defined for responders only, i.e. patients with a CR or PR. The actual dates the tumor scans were performed will be used for this calculation. DOR for patients who have not progressed or died at the time of analysis will be censored at the date of their last tumor assessment.
Progression-free survival (PFS) | From the date of study treatment start until the date of the first observed progression or date of death due to any cause, if death occurs before progression is documented (for a maximum duration of 36 months).
  Progression-free survival (PFS) is defined as the time (days) from start of study treatment to date of first observed disease progression (investigator's radiological or clinical assessment) or death due to any cause, if death occurs before progression is documented. The actual date that the tumor scan was performed will be used for this calculation. If a tumor assessment is performed over more than one day (e.g. scans for chest and abdomen done on different days for the same evaluation), the earliest date will be used for the calculation of PFS. For patients without documented radiological or clinical progression or death at the time of analysis, PFS will be censored at the last actual visit date of tumor evaluation.
Overall survival (OS) | From the date of study treatment start until the date of death due to any cause (for a maximum duration of 36 months).
  Overall survival (OS) is defined as the time from start of study treatment to death due to any cause. Patients alive at the date of data cut-off for analysis will be censored at the last date known to be alive. If a patient is lost to follow-up before any assessment after assignment to treatment, this patient will be censored at 1 day.
Safety and tolerability endpoints | Day 1 up to 90 days after last dose of study drug.
  Individual listings of adverse events will be provided. Treatment-related adverse events evaluated using the National Cancer Institute's Common Terminology Criteria for Adverse Events (version 5.0). Adverse events will be reported as absolute numbers (n) and relative frequencies (%). Visualization of the results will be presented with help of tables and diagrams.
Area under the concentration-time curve (AUC) | Day 1 up to the date of the last dose of study drug.
  The concentration-times courses of all analytes will be tabulated by dose level.
Maximum serum concentration (Cmax) of Clofarabine | Day 1 up to the date of the last dose of study drug.
  The concentration-times courses of all analytes will be tabulated by dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Shahrokh F. Shariat Prof. Dr., Professor, Principal Investigator — Department of Urology, Medical University of Viernna
Locations (1):
- Department of Urology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Foss FM, Parker T. A Phase I Dose-Escalation Study of Clofarabine in Patients with Relapsed or Refractory Low-Grade or Intermediate-Grade B-Cell or T-Cell Lymphoma. Oncologist. 2018 Apr;23(4):397-e30. doi: 10.1634/theoncologist.2017-0658. Epub 2018 Feb 7. PMID 29438091
- [Background] Kantarjian HM, Erba HP, Claxton D, Arellano M, Lyons RM, Kovascovics T, Gabrilove J, Craig M, Douer D, Maris M, Petersdorf S, Shami PJ, Yeager AM, Eckert S, Abichandani R, Faderl S. Phase II study of clofarabine monotherapy in previously untreated older adults with acute myeloid leukemia and unfavorable prognostic factors. J Clin Oncol. 2010 Feb 1;28(4):549-55. doi: 10.1200/JCO.2009.23.3130. Epub 2009 Dec 21. PMID 20026805
- [Background] Kantarjian HM, Gandhi V, Kozuch P, Faderl S, Giles F, Cortes J, O'Brien S, Ibrahim N, Khuri F, Du M, Rios MB, Jeha S, McLaughlin P, Plunkett W, Keating M. Phase I clinical and pharmacology study of clofarabine in patients with solid and hematologic cancers. J Clin Oncol. 2003 Mar 15;21(6):1167-73. doi: 10.1200/JCO.2003.04.031. PMID 12637486
- [Background] Zhenchuk A, Lotfi K, Juliusson G, Albertioni F. Mechanisms of anti-cancer action and pharmacology of clofarabine. Biochem Pharmacol. 2009 Dec 1;78(11):1351-9. doi: 10.1016/j.bcp.2009.06.094. Epub 2009 Jul 1. PMID 19576186
- [Background] Gutmann M, Ertl IE, Herek P, Vician P, Pirker C, Nossing C, Brettner R, Lemberger U, Grausenburger R, Batlogg K, Baumfried O, Prantl I, Singh N, Laukhtina E, Oszwald A, Wasinger G, Comperat E, Berger W, Shariat SF, Englinger B. Clofarabine Has a Superior Therapeutic Window as compared to Gemcitabine in Preclinical Bladder Cancer Models. Eur Urol Oncol. 2024 Dec;7(6):1166-1170. doi: 10.1016/j.euo.2024.05.001. Epub 2024 May 16. PMID 38755094
- [Background] Ertl IE, Lemberger U, Ilijazi D, Hassler MR, Bruchbacher A, Brettner R, Kronabitter H, Gutmann M, Vician P, Zeitler G, Koren A, Lardeau CH, Mohr T, Haitel A, Comperat E, Oszwald A, Wasinger G, Clozel T, Elemento O, Kubicek S, Berger W, Shariat SF. Molecular and Pharmacological Bladder Cancer Therapy Screening: Discovery of Clofarabine as a Highly Active Compound. Eur Urol. 2022 Sep;82(3):261-270. doi: 10.1016/j.eururo.2022.03.009. Epub 2022 Apr 4. PMID 35393162